CLINICAL TRIAL: NCT06297642
Title: A Phase Ib Clinical Trial of TQB2928 Injection Combined With Penpulimab in the Treatment of Patients With Advanced Malignant Tumors.
Brief Title: TQB2928 Injection Combined With Penpulimab in Treatment of Advanced Malignant Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the current status of the same target research and the company's overall layout in the field of tumors, the early termination was determined after full communication with the principal investigator of the group leader unit.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2928-AK105-Ib-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-01

CONDITIONS: Advanced Malignant Neoplasm
MeSH Terms: interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2928 injection + Penpulimab (Experimental): TQB2928 injection combined with Penpulimab, 21 days as a treatment cycle.
  Interventions: Drug: TQB2928 injection; Drug: Penpulimab

INTERVENTIONS:
Drug: TQB2928 injection — Anti-CD47 monoclonal antibody
Drug: Penpulimab — Humanized Monoclonal Antibody to Programmed Cell Death Protein 1 (PD-1)

SUMMARY:
This study will evaluate the safety and efficiency of TQB2928 injection combined with Penpulimab in the treatment of patients with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent;
* Age: ≥18 years old (when signing the informed consent form); Eastern Cooperative Oncology Group (ECOG) score: 0 or 2 point; The expected survival period exceeds 3 months;
* Subject population: Histologically and/or cytologically confirmed advanced malignancies, including lymphomas and solid tumors.
* Relapse or treatment failure after previous standard treatment, or intolerance to standard treatment and no other better treatment options：
* Adequate treatment with PD-1/PD-L1 (including monotherapy or combination) without remission or disease progression after treatment.
* Adequate main organs function
* Female subjects of childbearing age should agree to use contraceptives (such as Intrauterine device, contraceptives or condoms) during the study period and within 6 months after the end of the study; The serum or urine Pregnancy test was negative within 7 days before the study was included, and must be non-lactating subjects; Male participants should agree to use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Tumor disease and history:

  1. Nodular lymphocyte dominant Hodgkin's lymphoma or gray area lymphoma.
  2. The tumor involves the central nervous system.
  3. People with a history of hemophagocytic syndrome or who have been assessed by the investigator as being at suspected risk.
  4. Has experienced or currently suffers from other malignant tumors within 3 years.
* Previous anti-tumor therapy:

  1. Previous use of other similar drugs.
  2. received systemic antitumor drugs (including drugs under investigation) within 4 weeks prior to initial administration, or received Chimeric Antigen Receptor T-cell (CAR-T) Therapy or Autologous hematopoietic stem cell transplantation( auto-HSCT) within 3 months prior to initial administration.
  3. Previously received allogeneic hematopoietic stem cell transplantation (allo-HSCT).
  4. any major surgical procedure, chemotherapy and/or radiotherapy, immunotherapy, or targeted therapy within 4 weeks prior to initial dosing.
  5. Less than 5 drug half-lives between the first administration and the previous oral targeted therapy (calculated from the end time of the last therapy).
  6. Received within 2 weeks before the first administration of Chinese patent drugs (including compound cantharides capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Brucea oil injection/capsule, Xiaoaiping tablet/injection, cinobufagin capsule, etc.) approved by the National Drug Administration (NMPA) with anti-tumor indications.
* Concomitant diseases and medical history:

  1. Liver abnormalities:
  2. Abnormal kidney:
  3. Cardiovascular and cerebrovascular abnormalities:
  4. History of immune deficiency:
  5. Lung diseases:
  6. Active bacterial, fungal, or viral infections requiring systemic treatment.
  7. Subjects with a history of hemolytic anemia from any cause (including Evans syndrome) or a positive Coombs test within 3 months prior to initial dosing.
  8. A prior history of unexplained severe allergies, known to be allergic to monoclonal drugs or exogenous human immunoglobulins.
  9. with a serious or poorly controlled disease that, in the judgment of the investigator and sponsor, poses a serious risk to the safety of the subjects or affects the completion of the study.
  10. History of drug abuse or drug use.
* Live attenuated vaccines were administered within 4 weeks before the first dose or during the planned study period. Inactivated Corona Virus Disease 2019 (COVID-19) and influenza vaccines are allowed.
* Subjects with concomitant diseases that, in the judgment of the investigator, seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are not suitable for enrollment for other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Baseline up to 3 weeks
  The relevant adverse reactions occurred within the first cycle
Adverse event rate | Baseline up to 96 weeks
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Baseline up to 96 weeks
  Percentage of participants achieve complete response and partial response
Complete response rate (CRR) | Baseline up to 96 weeks
  Percentage of participants achieve complete response
Disease Control Rate | Baseline up to 96 weeks
  It is the proportion of patients whose tumors have shrunk or stabilized for a certain amount of time and includes complete response (CR), partial response (PR), and stable (SD) cases
Duration of Response | Baseline up to 96 weeks
  The time when the participants first achieved CR or PR to disease progression or death from any cause
Progression-free Survival | Baseline up to 96 weeks
  The period between the beginning of treatment and the observation of disease progression or death from any cause in a patient with a tumor disease
Overall survival (OS) | Baseline up to 96 weeks
  From the first injection to the time of death from any cause.
Incidence of Anti-Drug antibody | Cycle 1 day 1, Cycle 5 day 1, and 28 days, 90 days after the last administration. (Each cycle 21 days)
  The incidence of anti-drug antibody after administration of TQB2928 injection and penpulimab
Incidence of neutralizing antibodies | Cycle 1 day 1, Cycle 5 day 1, and 28 days, 90 days after the last administration. (Each cycle 21 days)
  The incidence of neutralizing antibodies after administration of TQB2928 injection and penpulimab
Peak time (Tmax) | Day 1, day 2 , day 4 , day 6 , day 8, day15 of cycle 1 and cycle 2. Each cycle 21 days.
  The time to peak concentration
Peak concentration (Cmax) | Day 1, day 2 , day 4 , day 6 , day 8, day15 of cycle 1 and cycle 2. Each cycle 21 days.
  Maximum plasma drug concentration
The area under the plasma concentration time curve from zero to after 24h (AUC0-24h) | Day 1, day 2 , day 4 , day 6 , day 8, day15 of cycle 1 and cycle 2. Each cycle 21 days.
  Area under the plasma concentration time curve from zero to after 24h for TQB2928.
Steady-state apparent volume of distribution (Vz/F) | Day 1, day 2 , day 4 , day 6 , day 8, day15 of cycle 1 and cycle 2. Each cycle 21 days.
  The total volume of body fluid required by the measured plasma drug concentration after the total amount of drug in the body is to be balanced.
Minimum plasma concentration at steady state (Cmin,ss) | Day 1, day 2 , day 4 , day 6 , day 8, day15 of cycle 1 and cycle 2. Each cycle 21 days.
  The minimum plasma concentration after stabilization
Receptor Occupancy (RO%) | day 1 and day 8 of Cycle 1, day 1 and day 15 of Cycle 2, 28 days after the last administration. (each cycle 21 days)
  The extent to which antibody drugs occupy cell surface targets

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Lu'an People's Hospital of Anhui Province, Lu'an, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong